CLINICAL TRIAL: NCT03352999
Title: Refractory Cardiac Arrest Management With Veno-Arterial Extra Corporeal Oxygenation Membrane Registry
Brief Title: Cardiac Arrest Extra Corporeal Oxygenation Membrane
Acronym: CAREECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A01873-48.
Record Dates: First submitted 2017-11-16; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Cardiac Arrest; Cardiopulmonary Resuscitation; Advanced Cardiac Life Support; Extracorporeal Life Support
Keywords: Refractory out-hospital cardiac arrest; Extracorporeal Life Support
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, open, routine care assessment study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ROHCA rescued by vaECMO (Other): Patients experiencing a ROHCA despite advanced CPR and finally rescued with a va ECMO device.
  Interventions: Procedure: Fast track access to vaECMO

INTERVENTIONS:
Procedure: Fast track access to vaECMO — ROHCA must be witnessed with onset of bystander CPR and an immediate call to Emergency Dispatch. Furthermore, to minimize any loss of time, all qualified geographical locations are directly incorporated in the regulation software of the center for medical emergency control.
  Patients suitable for vaECMO implantation were identified as early as possible by the Medical Dispatcher at the Emergency Call Dispatch Center.
  Bystanders pursued CPR until Mobile Intensive Care Unit (MICU) arrival. OHCA was considered refractory after 10 min of CPR initiating the transport by MICU to the hospital such that the vaECMO intervention could be performed. The resuscitation was pursued during the transfer to hospital. An automated chest compression device was used in order to minimize interruption periods.
  The intensivists and cardiac surgeons stood ready to implant the vaECMO surgically in the catheterization laboratory where a percutaneous coronary intervention was subsequently performed.

SUMMARY:
French guidelines for Cardio Pulmonary Resuscitation (CPR) consider Extra-Corporeal Life Support (ECLS) as one option in Refractory out-of hospital Cardiac Arrest (ROHCA) patients with a no-flow less than five minutes and absence of spontaneous circulation 30 minutes after initiation of advanced CPR. Duration of both pre-CPR arrest (no-flow) and of CPR (low-flow) have been systematically highlighted as crucial prognostic factors in all observational studies focused on ROHCA.

In order to shorten the time to ECLS initiation, the most recent European Resuscitation Council guidelines recommend, in eligible ROHCA patients, a fast track access to ECLS implantation.

CHRU Nancy elaborated an operational strategy which was designed to improve the enrolment of eligible ROHCA patients and to reduce the delay time between recognition and ECLS initiation.

The objective of the present register was to assess prospectively the impact of this new operational strategy over a 5 years period.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed out-of-hospital cardiac arrest
* in qualified geographical locations
* No Return of spontaneous circulation (ROSC) after 10 min of CPR
* No Flow <1 min

Exclusion Criteria:

* Apparent obvious comorbidities
* Patient < 18 yo
* Pregnancy
* Patient under protective supervision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of survivors without neurological sequelae Number of survivors without neurological sequelae (DRS scale from 0 to 6) | 1 year
  Number of survivors without neurological sequelae (DRS scale from 0 to 6)

SECONDARY OUTCOMES:
Number of survivors with or without neurological sequelae. | at 3 months
  Number of survivors with or without neurological sequelae (DRS from 0 to 29)
Number of survivors with or without neurological sequelae. | at 3 months
  European quality of life scale EQ-5D at 3 months
Ischemia-reperfusion assessment | from ECMO implantation and day 3
  Amount of fluid infused
Renal failure | ECMO implantation - Day 1- Day 3
  Worst KDIGO stage
Hepatic failure | ECMO implantation - Day 1 - Day 3
  Worst values of PT/bilirubin/ AST and ALT
Coagulation Failure | ECMO implantation- Day 1 - Day 3
  platelets/PT/Fibrinogen
Respiratory failure | ECMO implantation - Day 1- Day 3
  PaO2/iFO2 value
Hemodynamic Failure | from ECMO implantation and day 3
  Amount of Norepinephrine infused
Quality of Resuscitation | from collapse to ECMO implantation (up to 60 minutes)
  Total duration of the resuscitation: from collapse to ECMO implantation
Pupillary status | at arrival in intensive care - Hour 0 - Hour 6 - Hour 12 - Day 1
  Pupillary status
Lactate | Hour 0 - Hour 6 - Hour 12 - Day 1
  amount of Lactate
bispectral index | at arrival in intensive care - Hour 6 - Hour 12 - Day 1
  bispectral index
Nosocomial complications | ECMO implantation - Day 1 - Day 3
  Infection of the canulation site
Nosocomial complications | ECMO implantation - Day 1 - Day 3
  bacteraemia
Bleeding complications | ECMO implantation - Day 1 - Day 3
  blood hemostasis disorder
Bleeding complications | ECMO implantation - Day 1 - Day 3
  bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Kimmoun, MD, Principal Investigator — CHRU Nancy

REFERENCES:
- [Result] Chouihed T, Kimmoun A, Lauvray A, Laithier FX, Jaeger D, Lemoine S, Maureira JP, Nace L, Duarte K, Albizzati S, Girerd N, Levy B. Improving Patient Selection for Refractory Out of Hospital Cardiac Arrest Treated with Extracorporeal Life Support. Shock. 2018 Jan;49(1):24-28. doi: 10.1097/SHK.0000000000000941. PMID 28682938